CLINICAL TRIAL: NCT03875508
Title: Plaque Psoriasis: Usability of the Risankizumab Autoinjector Combination Product in Adults With Moderate to Severe Psoriasis
Brief Title: A Study to Assess Usability of Risankizumab Autoinjector Combination Product in Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-005
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Risankizumab; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Risankizumab (Experimental): Risankizumab solution (150 mg/mL) for injection; self-administered subcutaneously via a pre-filled autoinjector at Weeks 0, 4, 16, and 28
  Interventions: Drug: Risankizumab; Device: Autoinjector

INTERVENTIONS:
Drug: Risankizumab — Risankizumab to be injected subcutaneously (SC)
  Other Names: ABBV-066; BI 655066
Device: Autoinjector — Single dose pre-filled autoinjector containing risankizumab for SC injection

SUMMARY:
The objectives of this study were to evaluate the usability of the combination product of risankizumab in an autoinjector (AI), as well as to evaluate the efficacy, safety, and tolerability of risankizumab administered by AI for the treatment of adult participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This was a Phase 3 multicenter, single-arm, open-label study that evaluated usability and efficacy of the risankizumab-AI combination product. The study included a 30-day screening period with study visits at Weeks 0, 4, 16, 28, and 40 with a subsequent follow-up telephone call at approximately 20 weeks after the last dose of study drug (Week 48). Study drug dosing consisted of 4 self-administered doses given subcutaneously on Weeks 0, 4, 16, and 28. Dosing on Weeks 4 and 16 was self-administered at home.

ELIGIBILITY:
Inclusion Criteria:

* Participant has diagnosis of chronic plaque psoriasis for at least 6 months before the baseline visit
* Participant meets following disease activity criteria:

  * Stable moderate to severe chronic plaque psoriasis, defined as ≥ 10% body surface area (BSA) psoriasis involvement, static Physician Global Assessment (sPGA) score ≥ 3, and Psoriasis Area Severity Index (PASI) ≥ 12 at Screening and baseline visit
  * Candidate for systemic therapy as assessed by the investigator

Exclusion Criteria:

* Participant has history of active skin disease other than psoriasis that could interfere with the assessment of psoriasis
* Participant has history of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis
* Participant has previous exposure to risankizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (26):
- United States (26):
  - Advanced Research Associates /ID# 210634, Glendale, Arizona
  - Cognitive Clinical Trials /ID# 210770, Scottsdale, Arizona
  - Burke Pharmaceutical Research /ID# 211386, Hot Springs, Arkansas
  - Bakersfield Derma & Skin Cance /ID# 210773, Bakersfield, California
  - Encino Research Center / T. Jo /ID# 211735, Encino, California
  - Tien Q Nguyen MD, Inc /ID# 210775, Fountain Valley, California
  - UC Davis Health /ID# 210411, Sacramento, California
  - Dermatology Physicians of CT /ID# 210637, Shelton, Connecticut
  - Florida Academic Centers Research /ID# 210337, Coral Gables, Florida
  - Medallion Clinical Research Institute, LLC /ID# 210329, Naples, Florida
  - Renstar Medical Research /ID# 210878, Ocala, Florida
  - Epiphany Dermatology /ID# 211493, Overland Park, Kansas
  - DermAssociates /ID# 210838, Rockville, Maryland
  - Great Lakes Research, Inc. /ID# 210192, Bay City, Michigan
  - Somerset Skin Centre /ID# 211596, Troy, Michigan
  - Central Dermatology, PC /ID# 210301, St Louis, Missouri
  - AllCutis Research Inc /ID# 211429, Portsmouth, New Hampshire
  - Medication Management, LLC /ID# 213217, Greensboro, North Carolina
  - Oregon Medical Res Center PC /ID# 210334, Portland, Oregon
  - University of Pittsburgh MC /ID# 210839, Pittsburgh, Pennsylvania
  - Center for Clinical Studies /ID# 211565, Cypress, Texas
  - Center for Clinical Studies /ID# 210362, Houston, Texas
  - Suzanne Bruce and Associates /ID# 212210, Houston, Texas
  - Austin Institute for Clinical Research /ID# 212203, Pflugerville, Texas
  - Premier Clinical Research /ID# 212209, Spokane, Washington
  - Froedtert Mem Lutheran Hosp /ID# 210194, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat (ITT) population: all participants who received at least one dose of study drug
Period: Overall Study
Arm/Group | Risankizumab
Started | 108
Completed | 96
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 8
Not completed — Lack of Efficacy | 1
Not completed — Other, not specified | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants who received at least one dose of study drug
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95
  Black or African American | 5
  Asian | 7
  American Indian or Alaska Native | 1
  Native Hawaiian or other Pacific Islander | 0
  Other | 0
  Multiple | 0
  Missing | 0
Prior Use of Systemic Biologic for Psoriasis [Count of Participants; unit: Participants]
  0 | 60
  ≥1 | 48
Static Physician Global Assessment (sPGA) Score at Baseline [Count of Participants; unit: Participants] — The sPGA is an investigator assessment of the overall disease severity at the time of evaluation. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
  Participants
    Score of 3 | 88
    Score of 4 | 20
Psoriasis Area and Severity Index (PASI) Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
  units on a scale | 19.834 (7.2424)
Body Surface Area (BSA) Psoriasis Involvement at Baseline [Mean (Standard Deviation); unit: Percentage of body surface area affected] | 25.471 (17.4671)
Duration of Plaque Psoriasis [Mean (Standard Deviation); unit: years] | 16.89 (13.095)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Observer Rating of Successful Participant Self-administration
Description: Successful participant self-administration is defined as successfully completed the sequence of 4 critical steps in the Instructions for Use (IFU) without errors to administer study drug via the autoinjector. The steps are "chose an appropriate injection site"; "removed cap from autoinjector"; "activated the injection"; and "performed a complete injection".
Time Frame: Day 1 and Week 28
Population: Intent-to-treat (ITT) population: all participants who received at least one dose of study drug and had available data
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 104
percentage of participants
  Day 1 | 100
  Week 28: number analyzed (Participants) | 98
  Week 28 | 100

2. Primary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 90 at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at Week 16) / PASI score at Baseline * 100.
Time Frame: At Week 16
Population: Intent-to-treat (ITT) population: all participants who received at least one dose of study drug; those with missing data were imputed as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
percentage of participants | 66.7 [57.8 to 75.6]

3. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of Clear or Almost Clear at Week 16
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
percentage of participants | 81.5 [74.2 to 88.8]

4. Primary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 100 at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at Week 16) / PASI score at Baseline * 100.
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
percentage of participants | 46.3 [36.9 to 55.7]

5. Primary Outcome: Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at Week 16) / PASI score at Baseline * 100.
Time Frame: At Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
percentage of participants | 84.3 [77.4 to 91.1]

6. Primary Outcome: Percentage of Participants Who Had No Potential Hazards as Measured by an Observer
Description: Potential hazards are measured by an observer on the possible use-related hazards checklist for self-administration with the autoinjector. Hazards include injection at incorrect site; administration delayed because of cap removal difficulties; slip hazard during cap disposal attempt; small component swallowed after incorrect disposal of cap; patient received less medication than intended; needle shield did not deploy and resulted in sharps exposure; and pen not discarded properly and resulted in a biohazard for others.
Time Frame: Day 1 and Week 28
Population: Intent-to-treat (ITT) population: all participants who received at least one dose of study drug and had available data
Measure: Number; unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 103
percentage of participants
  Day 1 | 100
  Week 28: number analyzed (Participants) | 98
  Week 28 | 100

7. Primary Outcome: Participant Rating of Acceptability by the Self-Injection Assessment Questionnaire (SIAQ)
Description: Participants completed the Self-Injection Assessment Questionnaire (SIAQ), an instrument previously validated in those with rheumatoid arthritis, on an electronic patient-report outcome (ePRO) device. The POST module includes four principal causal domains: feelings about injections, self-confidence, pain and reaction during or after the injection, and ease of use, plus two additional domains on satisfaction with self-injection and self-image. Participants rate each item of the SIAQ 20 to 40 minutes following injections, and the ratings are transformed to scores ranging from 0 (worst experience) to 10 (best experience). The domain score is the mean of the item scores included in the domain. Higher domain scores indicate wider acceptability by subjects to use the autoinjector.
Time Frame: Day 1, Week 4, Week 16, Week 28
Population: Intent-to-treat (ITT) population: all participants who received at least one dose of study drug and had available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 101
units on a scale
  Feelings about injections- Day 1 | 8.358 (2.3613)
  Self-confidence- Day 1 | 8.556 (2.0646)
  Satisfaction with self-injection- Day 1 | 9.056 (1.0321)
  Injection-site reactions- Day 1 | 9.817 (0.4469)
  Ease of use- Day 1 | 8.82 (1.415)
  Self-image- Day 1 | 9.53 (1.261)
  Feelings about injections- Week 4: number analyzed (Participants) | 98
  Feelings about injections- Week 4 | 8.478 (2.0024)
  Self-confidence- Week 4: number analyzed (Participants) | 98
  Self-confidence- Week 4 | 8.112 (2.6313)
  Satisfaction with self-injection- Week 4: number analyzed (Participants) | 98
  Satisfaction with self-injection- Week 4 | 9.096 (1.1572)
  Injection-site reactions- Week 4: number analyzed (Participants) | 98
  Injection-site reactions- Week 4 | 9.700 (0.5710)
  Ease of use- Week 4: number analyzed (Participants) | 98
  Ease of use- Week 4 | 8.84 (1.240)
  Self-image- Week 4: number analyzed (Participants) | 98
  Self-image- Week 4 | 9.16 (1.964)
  Feelings about injections- Week 16: number analyzed (Participants) | 100
  Feelings about injections- Week 16 | 8.750 (1.8483)
  Self-confidence- Week 16: number analyzed (Participants) | 100
  Self-confidence- Week 16 | 8.367 (2.5921)
  Satisfaction with self-injection- Week 16: number analyzed (Participants) | 100
  Satisfaction with self-injection- Week 16 | 9.229 (1.1517)
  Injection-site reactions- Week 16: number analyzed (Participants) | 100
  Injection-site reactions- Week 16 | 9.763 (0.4576)
  Ease of use- Week 16: number analyzed (Participants) | 100
  Ease of use- Week 16 | 8.93 (1.394)
  Self-image- Week 16: number analyzed (Participants) | 100
  Self-image- Week 16 | 9.28 (1.678)
  Feelings about injections- Week 28: number analyzed (Participants) | 83
  Feelings about injections- Week 28 | 8.675 (2.0661)
  Self-confidence- Week 28: number analyzed (Participants) | 83
  Self-confidence- Week 28 | 8.795 (2.3034)
  Satisfaction with self-injection- Week 28: number analyzed (Participants) | 83
  Satisfaction with self-injection- Week 28 | 9.458 (1.0500)
  Injection-site reactions- Week 28: number analyzed (Participants) | 83
  Injection-site reactions- Week 28 | 9.725 (0.8911)
  Ease of use- Week 28: number analyzed (Participants) | 83
  Ease of use- Week 28 | 9.39 (0.971)
  Self-image- Week 28: number analyzed (Participants) | 83
  Self-image- Week 28 | 9.34 (1.614)

8. Other Pre Specified Outcome: Percent Change From Baseline in Psoriasis Area Severity Index (PASI) Score up to Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked.The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. Negative values indicate an improvement from baseline.
Time Frame: Baseline, Week 4, and Week 16
Population: Intent-to-treat (ITT) population: all randomized participants with a non-missing baseline measurement and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from Baseline
Arm/Group | Risankizumab
Number analyzed (Participants) | 107
percent change from Baseline
  Week 4 | -61.57 [-66.502 to -56.636]
  Week 16: number analyzed (Participants) | 106
  Week 16 | -89.33 [-92.915 to -85.750]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 20 weeks after last study drug administration, up to 48 weeks. In addition, serious adverse events and protocol-related nonserious adverse events were collected from the time the participant signed the study-specific informed consent.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 20 weeks have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 6/108
Other Adverse Events (participants affected / at risk) | 12/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=108)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=108)
NASOPHARYNGITIS (Infections and infestations) | 8 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03875508/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03875508/SAP_001.pdf